CLINICAL TRIAL: NCT03343054
Title: A PHASE 1 STUDY OF THE SAFETY, PHARMACOKINETICS AND ANTI-TUMOR ACTIVITY OF TALAZOPARIB, POLY (ADP-RIBOSE) POLYMERASE (PARP) INHIBITOR, IN JAPANESE PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: A Phase 1 Study Of Talazoparib, PARP Inhibitor, In Japanese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3441030
Record Dates: First submitted 2017-11-11; First posted 2017-11-17 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Neoplasms; Breast Neoplasms
Keywords: Phase 1; talazoparib; PF-06944076; MDV3800; BMN673; PARP inhibitor; Japanese; solid tumors; breast cancer; C3441030
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- talazoparib (Experimental): 0.75 mg/day or 1.0 mg/day
  Interventions: Drug: talazoparib

INTERVENTIONS:
Drug: talazoparib — Talazoparib will be administered orally on a continuous basis. Talazoparib may be taken with or without food. Each cycle will consist of 28 days.

SUMMARY:
This is a Phase 1 study which consists of 2 parts; Dose Escalation part and Expansion part.

The dose escalation part is open-label, and evaluates safety, preliminary efficacy and PK of single-agent talazoparib in sequential cohorts of adult patients with advanced solid tumors who are resistant to standard therapy or for whom no standard therapy is available.

In the dose escalation part, up to 18 (minimum 3) patients are expected to be enrolled depending on the observed DLTs.

The expansion part is designed to assess the efficacy, safety and PK of single-agent talazoparib at RP2D determined in the dose escalation part in adult patients with locally advanced or metastatic breast cancer who have deleterious or suspected deleterious germline BRCA1 or BRCA2 mutations.

In the expansion part, a minimum of 17 patients will be enrolled evaluable for the primary endpoint.

ELIGIBILITY:
[Dose Escalation Part]

Inclusion Criteria:

* Histological or cytological diagnosis of locally advanced or metastatic solid tumor that is resistant to standard therapy or for which no standard therapy is available.
* ECOG Performance Status 0 or 1.
* Adequate Bone Marrow, Renal and Liver Function.

Exclusion Criteria:

* Patients with known symptomatic brain metastases requiring steroids.
* Current use of a strong P-gp inhibitor, strong P-gp inducer, or strong inhibitor of BCRP within 1 week or 5 half lives which ever is longer prior to the first dose of study treatment.
* Fertile male patients and female patients of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception.

[Dose Expansion Part]

Inclusion Criteria:

* Histologically or cytologically confirmed carcinoma of the breast.
* Locally advanced breast cancer that is not amenable to curative radiation or surgery and/or metastatic disease.
* Documentation of a deleterious, suspected deleterious, or pathogenic germline BRCA1 or BRCA2 mutation by Myriad Genetics' BRACAnalysis CDx test.
* No more than 3 prior chemotherapy-inclusive regimens for locally advanced or metastatic disease.
* Have measurable lesion by the RECIST v.1.1.
* ECOG Performance Status 0-2.
* Adequate Bone Marrow, Renal and Liver Function.

Exclusion Criteria:

* First-line locally advanced or metastatic breast cancer with no prior neoadjuvant and adjuvant chemotherapy.
* Prior treatment with a PARP inhibitor.
* Objective disease progression while receiving platinum chemotherapy administered for locally advanced or metastatic disease.
* HER2 positive breast cancer.
* Active inflammatory breast cancer.
* Central nervous system (CNS) metastases.
* Current or anticipated use within 7 days prior to the first dose of study treatment, or anticipated use during the study of strong P-gp inhibitors.
* Fertile male patients and female patients of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2024-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Japan (8):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima
  - National Hospital Organization Osaka National Hospital, Osaka

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Kotani H, Masuda N, Yamashita T, Naito Y, Taira T, Inoue K, Takahashi M, Yonemori K, Toyoizumi S, Mori Y, Nagasawa T, Hori N, Iwata H. Efficacy and safety of talazoparib in Japanese patients with germline BRCA-mutated locally advanced or metastatic breast cancer: results of the phase 1 dose-expansion study. Breast Cancer. 2022 Nov;29(6):1088-1098. doi: 10.1007/s12282-022-01390-w. Epub 2022 Jul 30. PMID 35907135
- [Derived] Naito Y, Kuboki Y, Ikeda M, Harano K, Matsubara N, Toyoizumi S, Mori Y, Hori N, Nagasawa T, Kogawa T. Safety, pharmacokinetics, and preliminary efficacy of the PARP inhibitor talazoparib in Japanese patients with advanced solid tumors: phase 1 study. Invest New Drugs. 2021 Dec;39(6):1568-1576. doi: 10.1007/s10637-021-01120-7. Epub 2021 Jun 23. PMID 34160752
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included 2 periods: dose escalation and dose expansion. The recommended dose for dose expansion period of talazoparib was determined in dose escalation period.
Pre-assignment Details: Dose escalation period: total 9 participants were screened, enrolled into the study and assigned to study treatment. Dose expansion period: total 22 participants were screened, out of which 3 participants were screen failure. 19 participants actually enrolled into the study and assigned to study treatment. Data reported based on the primary completion date of 11 January 2021.
Groups:
- Dose Escalation: Talazoparib 0.75 mg: Participants with advanced solid tumors who were resistant to standard therapy or for whom no standard therapy was available, received talazoparib capsules at a dose of 0.75 milligrams (mg) orally, once daily (QD) in each 28-day treatment cycle (except Cycle 1 with 7 additional days lead-in) until disease progression, unacceptable toxicity or withdrawal of consent (maximum duration: up to 286 days). Cycle 1 contained a 7 day lead-in phase in which participants received single dose of 0.75 mg talazoparib on Day minus (-) 7.
- Dose Escalation: Talazoparib 1.0 mg: Participants with advanced solid tumors who were resistant to standard therapy or for whom no standard therapy was available, received talazoparib capsules at a dose of 1.0 mg orally QD in each 28-day treatment cycle (except Cycle 1 with 7 additional days lead-in) until disease progression, unacceptable toxicity or withdrawal of consent (maximum duration: up to 286 days). Cycle 1 contained a 7 day lead-in phase in which participants received single dose of 1.0 mg talazoparib on Day -7.
- Dose Expansion: Talazoparib 1.0 mg: Participants with Germline breast cancer susceptibility gene mutation (gBRCAm) HER2-negative locally advanced or metastatic breast cancer, received talazoparib capsules at a dose of 1.0 mg orally QD in each 28-day treatment cycle until disease progression, unacceptable toxicity or withdrawal of consent (maximum duration: up to 502 days).
Period: Dose Escalation Period (Up to 286 Days)
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg | Dose Expansion: Talazoparib 1.0 mg
Started | 3 | 6 | 0 (Dose escalation and Dose expansion were separate populations.)
Completed | 0 | 0 | 0
Not Completed | 3 | 6 | 0
Not completed — Progressive Disease | 2 | 6 | 0
Not completed — Global Deterioration of Health Status | 1 | 0 | 0
Period: Dose Expansion Period (Up to 502 Days)
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg | Dose Expansion: Talazoparib 1.0 mg
Started | 0 | 0 | 19 (Dose escalation and Dose expansion were separate populations.)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 19
Not completed — Progressive Disease | 0 | 0 | 11
Not completed — Ongoing | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants assigned to study treatment and who took at least 1 dose of study treatment.
Groups:
- Dose Escalation: Talazoparib 0.75 mg: Participants with advanced solid tumors who were resistant to standard therapy or for whom no standard therapy was available, received talazoparib capsules at a dose of 0.75 mg orally, QD in each 28-day treatment cycle (except Cycle 1 with 7 additional days lead-in) until disease progression, unacceptable toxicity or withdrawal of consent (maximum duration: up to 286 days). Cycle 1 contained a 7 day lead-in phase in which participants received single dose of 0.75 mg talazoparib on Day -7.
- Dose Expansion: Talazoparib 1.0 mg: Participants with gBRCAm HER2-negative locally advanced or metastatic breast cancer, received talazoparib capsules at a dose of 1.0 mg orally QD in each 28-day treatment cycle until disease progression, unacceptable toxicity or withdrawal of consent (maximum duration: up to 502 days).
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg | Dose Expansion: Talazoparib 1.0 mg | Total
Number analyzed (Participants) | 3 | 6 | 19 | 28
Age, Customized [Count of Participants; unit: Participants]
  Less than (<)18 Years | 0 | 0 | 0 | 0
  18-44 Years | 1 | 0 | 7 | 8
  45-64 Years | 1 | 3 | 6 | 10
  Greater than or equal to (>=)65 Years | 1 | 3 | 6 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 19 | 24
  Male | 1 | 3 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 19 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 6 | 19 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: DLT was defined as any of the following adverse events occurred in 1st treatment cycle and attributable to talazoparib: hematologic- grade(G) 4 neutropenia greater than (>)7days; Febrile neutropenia >1 hour; G greater than or equal to (>=)3 neutropenic infection, thrombocytopenia associated with G2 hemorrhage; G4 thrombocytopenia, anemia; G3 anemia required transfusion; daily dosing interrupted for >=7 total days in first cycle for G3 neutropenia/thrombocytopenia. Non-hematologic: any G>=3AE except non-clinically significant laboratory abnormalities, Non-hematologic AE deemed not clinically significant, nausea, vomiting, diarrhea responded to medical intervention within 72 hours, fatigue improved to G>=2 within 7 days. Alanine/aspartate aminotransferase (ALT/AST)>5*upper limit of normal(ULN) and 2*increases above baseline values; ALT/AST>=3*ULN concurrent with total bilirubin (TB)>2*ULN; TB>5*ULN; failure to deliver 75percent(%) of doses due to toxicities attributable to talazoparib.
Time Frame: Cycle 1 (28 days)
Population: The per-protocol analysis set included all enrolled participants who received at least 1 dose of study treatment and who did not have major treatment deviations during the first cycle. Data for this outcome measure was not planned to be collected and analyzed for dose expansion period.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

2. Primary Outcome: Dose Expansion: Percentage of Participants With Confirmed Objective Response (OR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 by Investigator Assessment
Description: Confirmed OR in participants was defined as the percentage of participants with complete response (CR) or partial response (PR) as best response determined by investigator as per RECIST v 1.1 and confirmed by a second image at least 4 weeks from the initial imaging showing response. As per RECIST v 1.1, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From start of the treatment until disease progression or death (due to any cause) whichever occurred first (maximum duration: up to 502 days)
Population: FAS included all participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 19
Percentage of participants | 57.9 [36.8 to 77.0]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) Based on National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.03
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event was the AE resulting in any of following outcomes/deemed significant for any other reason: death; initial /prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were the events between first dose of study drug and up to 30 days after last dose or before start of new anticancer therapy, whichever occurred first. TEAE graded by CTCAE v 4.03 as Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death.
Time Frame: From start of the treatment up to 30 days after last dose or start of new anticancer therapy, whichever occurred first (Dose escalation: maximum duration- up to 286 days; Dose expansion: maximum duration- up to 502 days)
Population: The safety analysis set (SAS) included all participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6 | 19
Participants | 3 | 6 | 19

4. Secondary Outcome: Number of Participants With Treatment Related Adverse Events Based on National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.03
Description: A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. Serious adverse event was the AE resulting in any of following outcomes/deemed significant for any other reason: death; initial /prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were the events between first dose of study drug and up to 30 days after last dose or before start of new anticancer therapy, whichever occurred first. AE graded by CTCAE v 4.03 as Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death. Relatedness to study drug was assessed by the investigator.
Time Frame: as for outcome 3
Population: The safety analysis set included all participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6 | 19
Participants | 2 | 3 | 19

5. Secondary Outcome: Number of Participants With Grade 3 or Higher Treatment-Emergent Adverse Events (AEs) Based on National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.03
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were the events between first dose of study drug and up to 30 days after last dose or before start of new anticancer therapy, whichever occurred first. TEAE graded by CTCAE v 4.03 as Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death. In this outcome measure, number of participants with grade 3 or higher AEs were reported.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6 | 19
Participants | 1 | 2 | 11

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities Based on National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.03: Chemistry
Description: Parameters: Alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, creatinine increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, hypophosphatemia. As per CTCAE v 4.03: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening. Only those categories in which at least one participant had data were reported in this outcome measure.
Time Frame: Dose escalation: Baseline up to 286 days; Dose expansion: Baseline up to 502 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6 | 19
Participants
  Alanine aminotransferase increased: Grade 1 | 1 | 2 | 8
  Alanine aminotransferase increased: Grade 2 | 0 | 0 | 1
  Alkaline phosphatase increased: Grade 1 | 1 | 2 | 4
  Alkaline phosphatase increased: Grade 2 | 0 | 1 | 1
  Aspartate aminotransferase increased: Grade 1 | 1 | 3 | 7
  Blood bilirubin increased: Grade 1 | 0 | 0 | 2
  Creatinine increased: Grade 1 | 2 | 6 | 17
  Hyperglycemia: Grade 1 | 0 | 0 | 1
  Hyperkalemia: Grade 1 | 1 | 0 | 0
  Hypermagnesemia: Grade 1 | 0 | 0 | 1
  Hypernatremia: Grade 1 | 0 | 1 | 1
  Hypoalbuminemia: Grade 1 | 2 | 2 | 6
  Hypoalbuminemia: Grade 2 | 0 | 1 | 0
  Hypocalcemia: Grade 1 | 1 | 2 | 9
  Hypoglycemia: Grade 1 | 0 | 0 | 1
  Hypomagnesemia: Grade 1 | 0 | 1 | 2
  Hyponatremia: Grade 1 | 1 | 1 | 2
  Hypophosphatemia: Grade 2 | 1 | 1 | 2

7. Secondary Outcome: Number of Participants With Laboratory Abnormalities Based on National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.03: Hematology
Description: Hematological parameters included: Anemia, Hemoglobin increased, Lymphocyte count decreased, Lymphocyte count increased, Neutrophil count decreased, Platelet count decreased, White blood cell decreased. As per CTCAE v 4.03: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening. Only those categories in which at least one participant had data were reported in this outcome measure.
Time Frame: Dose escalation: Baseline up to 286 days; Dose expansion: Baseline up to 502 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6 | 19
Participants
  Anemia: Grade 1 | 3 | 2 | 8
  Anemia: Grade 2 | 0 | 3 | 0
  Anemia: Grade 3 | 0 | 1 | 9
  Lymphocyte count decreased: Grade 1 | 1 | 2 | 6
  Lymphocyte count decreased: Grade 2 | 2 | 3 | 4
  Lymphocyte count decreased: Grade 3 | 0 | 1 | 2
  Neutrophil count decreased: Grade 2 | 1 | 0 | 7
  Neutrophil count decreased: Grade 3 | 0 | 1 | 4
  Platelet count decreased: Grade 1 | 1 | 1 | 10
  Platelet count decreased: Grade 2 | 0 | 1 | 1
  White blood cell decreased: Grade 1 | 1 | 2 | 1
  White blood cell decreased: Grade 2 | 1 | 1 | 9
  White blood cell decreased: Grade 3 | 0 | 1 | 2

8. Secondary Outcome: Dose Escalation: Number of Participants With Abnormalities in Vital Signs
Description: Vital sign abnormalities: a) Sitting systolic blood pressure: <90 millimeter of mercury (mmHg), decrease from baseline >=30 mmHg, increase from baseline >=30 mmHg; b) Sitting diastolic blood pressure: minimum <50 mmHg, decrease from baseline >=20 mmHg, increase from baseline >=20 mmHg; c) Sitting pulse rate: minimum <40 beats per minute (bpm), maximum >120 bpm. Only those categories in which at least one participant had data were reported in this outcome measure.
Time Frame: Baseline up to 286 days
Population: The safety analysis set included all participants assigned to study treatment and who took at least 1 dose of study treatment. Data for this outcome measure was not planned to be collected and analyzed for dose expansion period, as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Participants
  Systolic blood pressure: <90 mmHg | 1 | 0
  Systolic blood pressure: decrease from baseline >=30 mmHg | 0 | 2

9. Secondary Outcome: Dose Escalation- Single Dose: Maximum Observed Plasma Concentration (Cmax) for Talazoparib
Description: Cmax was defined as the maximum observed plasma concentration of talazoparib.
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post dose on Day -7 of Cycle 1
Population: The Pharmacokinetic (PK) parameter analysis set included all enrolled participants treated who had sufficient information to estimate at least 1 of the pharmacokinetic parameters of interest in the dose escalation period only. Data for this outcome measure was not planned to be collected and analyzed for dose expansion period, as pre-specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Nanogram per milliliter | 7.244 (34) | 13.78 (26)

10. Secondary Outcome: Dose Escalation- Single Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Talazoparib
Description: Tmax was defined as the time to reach maximum observed plasma concentration of talazoparib.
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post dose on Day -7 of Cycle 1
Population: The PK parameter analysis set included all enrolled participants treated who had sufficient information to estimate at least 1 of the pharmacokinetic parameters of interest in the dose escalation period only. Data for this outcome measure was not planned to be collected and analyzed for dose expansion period, as pre-specified in protocol.
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Hours | 0.983 [0.750 to 1.92] | 0.967 [0.467 to 1.98]

11. Secondary Outcome: Dose Escalation- Single Dose: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Talazoparib
Description: Area under the plasma concentration time-curve from time zero to the time of last measured concentration (AUClast).
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post dose on Day -7 of Cycle 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram hour per milliliter
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Nanogram hour per milliliter | 97.48 (17) | 159.1 (33)

12. Secondary Outcome: Dose Escalation- Single Dose: Area Under the Curve From Time Zero to Time Tau (AUCtau) for Talazoparib
Description: Area under the plasma concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 24 hours.
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10 and 24 hours post dose on Day -7 of Cycle 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram hour per milliliter
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Nanogram hour per milliliter | 46.55 (20) | 85.39 (44)

13. Secondary Outcome: Dose Escalation- Single Dose: Apparent Oral Clearance of Talazoparib (CL/F)
Description: Clearance is a measure of the rate at which a drug was metabolized or eliminated by normal biological processes.
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post dose on Day -7 of Cycle 1
Population: The PK parameter analysis set included all enrolled participants treated who had sufficient information to estimate at least 1 of the pharmacokinetic parameters of interest in the dose escalation period only. Here "overall number of participants analyzed" signifies participants evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for dose expansion period, as pre-specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 4
Liter per hour | 6.968 (12) | 5.010 (9)

14. Secondary Outcome: Dose Escalation- Single Dose: Apparent Volume of Distribution (Vz/F) for Talazoparib
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post dose on Day -7 of Cycle 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 4
Liter | 551.8 (42) | 361.1 (20)

15. Secondary Outcome: Dose Escalation- Single Dose: Terminal Half-Life (t1/2) for Talazoparib
Description: Terminal half-life (t1/2) is the time measured for the plasma concentration of a drug to decrease by half of its initial concentration.
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post dose on Day -7 of Cycle 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 4
Hours | 56.60 (17.860) | 50.73 (10.121)

16. Secondary Outcome: Dose Escalation- Single Dose: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for Talazoparib
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre dose) to extrapolated infinite time (0-inf).
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post dose on Day -7 of Cycle 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram hour per milliliter
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 4
Nanogram hour per milliliter | 107.5 (12) | 199.7 (9)

17. Secondary Outcome: Dose Escalation- Multiple Dose: Maximum Observed Plasma Concentration at Steady State (Css,Max) for Talazoparib
Description: Css,max is maximum observed plasma concentration at steady state (post multiple dose) of Talazoparib.
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10 and 24 hours post dose on Day 22 of Cycle 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Nanogram per milliliter | 14.44 (26) | 32.84 (14)

18. Secondary Outcome: Dose Escalation- Multiple Dose: Predose Concentration (Cmin) for Talazoparib
Description: Pre dose plasma concentration of talazoparib.
Time Frame: Pre dose on Day 22 of Cycle 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Nanogram per milliliter | 2.175 (8) | 3.645 (49)

19. Secondary Outcome: Dose Escalation- Multiple Dose: Time for Maximum Observed Plasma Concentration at Steady State (Tss,Max) for Talazoparib
Description: Tss,max = Time to reach Cmax for talazoparib at steady state (post multiple dose).
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10 and 24 hours post dose on Day 22 of Cycle 1
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Hours | 1.02 [0.967 to 1.87] | 1.03 [0.733 to 1.92]

20. Secondary Outcome: Dose Escalation- Multiple Dose: Area Under the Curve From Time Zero to Time Tau at Steady State (AUCss,Tau) for Talazoparib
Description: Area under the plasma concentration curve from time 0 to end of dosing interval (AUCtau) at steady state (post multiple dose), where dosing interval was 24 hours.
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10 and 24 hours post dose on Day 22 of Cycle 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram hour per milliliter
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Nanogram hour per milliliter | 127.2 (6) | 244.7 (21)

21. Secondary Outcome: Dose Escalation- Multiple Dose: Apparent Oral Clearance of Talazoparib at Steady State (CL/Fss)
Description: Clearance is a measure of the rate at which a drug was metabolized or eliminated by normal biological processes.
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10 and 24 hours post dose on Day 22 of Cycle 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Liter per hour | 5.898 (7) | 4.086 (21)

22. Secondary Outcome: Dose Escalation- Multiple Dose: Accumulation Ratio (Rac) of AUCtau for Talazoparib
Description: Accumulation ratio for AUC was calculated as AUCtau for Day 22 divided by AUCtau for Day -7, where AUCtau was defined as area under the plasma concentration curve from time 0 to end of dosing interval, where dosing interval was 24 hours.
Time Frame: Pre dose, 0.5, 0.75, 1, 2, 4, 6, 8, 10 and 24 hours post dose on Day -7 and Day 22 of Cycle 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Ratio | 2.734 (24) | 2.866 (64)

23. Secondary Outcome: Dose Escalation- Multiple Dose: Linearity Ratio (Rss) of AUC for Talazoparib
Description: Rss was calculated by dividing AUCtau at steady state (post multiple dosing on Day 22) by single dose AUCinf (on Day -7). AUCtau was defined as area under the plasma concentration curve from time 0 to end of dosing interval, where dosing interval was 24 hours. AUCinf was defined as area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: Pre dose, 0.50, 0.75, 1, 2, 3, 4, 6, 8, 10, 24, 48, 72 and 96 hours post dose on Day -7 of Cycle 1; Pre dose, 0.5, 0.75, 1, 2, 4, 6, 8, 10 and 24 hours post dose on Day 22 of Cycle 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 4
Ratio | 1.181 (12) | 1.249 (14)

24. Secondary Outcome: Dose Escalation: Percentage of Participants With Objective Response (OR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: OR in participants was defined as the percentage of participants with CR or PR as best response determined by investigator as per RECIST v 1.1. As per RECIST v 1.1, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From start of the treatment until disease progression or death (due to any cause) whichever occurred first (maximum duration: up to 286 days)
Population: FAS included all participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Percentage of participants | 0 | 0

25. Secondary Outcome: Dose Escalation: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of first dose of study drug to the earliest date of disease progression per RECIST v 1.1, or death due to any cause, whichever occurs first. PD = at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) and an absolute increase of >=5 mm or appearance of at least 1 new lesion.
Time Frame: From day of first dose until disease progression or death (due to any cause) whichever occur first (maximum duration: up to 286 days)
Population: FAS included all participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 3 | 6
Months | 3.0 [2.1 to 3.0] | 3.4 [1.2 to 9.6]

26. Secondary Outcome: Dose Escalation: Duration of Response (DOR)
Description: DOR was defined as the time between the date of the first documented objective response (PR or CR) and the date of the first documented progression or death (due to any cause) whichever occurs first. As per RECIST v 1.1: CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: From date of first documented response to date of first documented PD or death (due to any cause) whichever occurred first (maximum duration: up to 286 days)
Population: Due to no participants with response in dose escalation period, data collection and analysis for DOR was not performed. Hence, data is not reported.
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Dose Expansion: Percentage of Participants With Confirmed Objective Response (OR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Blinded Independent Central Review (BICR)
Description: Confirmed OR in participants was defined as the percentage of participants with CR or PR as best response determined by BICR as per RECIST v 1.1 and confirmed by a second image at least 4 weeks from the initial imaging showing response. As per RECIST v 1.1, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 2
Population: FAS included all participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 19
Percentage of participants | 52.6 [32.0 to 72.6]

28. Secondary Outcome: Dose Expansion: Percentage of Participants With Confirmed Disease Control as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Investigator Assessment
Description: Disease Control (DC) was defined as participants with a confirmed CR, confirmed PR and SD at 16 and 24 weeks as assessed by investigator as per RECIST v 1.1. As per RECIST v 1.1, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least a 20% increase in the sum of diameters of target lesions) taking as reference the smallest sum diameters while on study.
Time Frame: Baseline up to Week 16, Baseline up to Week 24
Population: FAS included all participants assigned to study treatment and who took at least 1 dose of study treatment. Data for this outcome measure was not planned to be collected and analyzed for dose escalation period, as pre-specified in protocol.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 19
Percentage of participants
  Up to Week 16 | 94.7 [77.4 to 99.7]
  Up to Week 24 | 94.7 [77.4 to 99.7]

29. Secondary Outcome: Dose Expansion: Percentage of Participants With Confirmed Disease Control as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Blinded Independent Central Review (BICR)
Description: Disease Control (DC) was defined as participants with a confirmed CR, confirmed PR and SD at 16 and 24 weeks as assessed by BICR as per RECIST v 1.1. As per RECIST v 1.1, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least a 20% increase in the sum of diameters of target lesions) taking as reference the smallest sum diameters while on study.
Time Frame: Baseline up to Week 16, Baseline up to Week 24
Population: as for outcome 28
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 19
Percentage of participants
  Up to Week 16 | 89.5 [70.4 to 98.1]
  Up to Week 24 | 89.5 [70.4 to 98.1]

30. Secondary Outcome: Dose Expansion: Time-to-Tumor Response (TTR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Investigator Assessment
Description: TTR was defined as the time (in months) from the date of first dose of study drug to the first documentation of objective response (CR or PR) as assessed by investigator according to RECIST v 1.1. As per RECIST v 1.1, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study drug until first documentation of CR or PR (maximum duration: up to 502 days)
Population: Analysis was performed on subset of participants with OR. Data for this outcome measure was not planned to be collected and analyzed for dose escalation period, as pre-specified in protocol.
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 11
Months | 2.63 [1.2 to 9.4]

31. Secondary Outcome: Dose Expansion: Time-to-Tumor Response (TTR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Blinded Independent Central Review (BICR)
Description: TTR was defined as the time (in months) from the date of first dose of study drug to the first documentation of objective response (CR or PR) as assessed by BICR according to RECIST v 1.1. As per RECIST v 1.1, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study drug until first documentation of CR or PR (maximum duration: up to 502 days)
Population: as for outcome 30
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 10
Months | 2.07 [1.2 to 4.2]

32. Secondary Outcome: Dose Expansion: Duration of Response (DOR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Investigator Assessment
Description: DOR was defined as the time between the date of first documented objective response (PR or CR) and the date of first documented progression or death (due to any cause) whichever occurs first. As per RECIST v 1.1: CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: From date of first documented response to date of first documented PD or death (due to any cause) whichever occurred first (maximum duration: up to 502 days)
Population: Analysis was performed on subset of participants with OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 11
Months | 6.8 [2.7 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to low number of participants with event.

33. Secondary Outcome: Dose Expansion: Duration of Response (DOR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Blinded Independent Central Review (BICR)
Description: as for outcome 32
Time Frame: as for outcome 32
Population: Analysis was performed on subset of participants with OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 10
Months | 6.0 [2.3 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with event.

34. Secondary Outcome: Dose Expansion: Progression Free Survival (PFS) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Investigator Assessment
Description: as for outcome 25
Time Frame: From day of first dose until disease progression or death (due to any cause) whichever occur first (maximum duration: up to 502 days)
Population: FAS included all participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 19
Months | 7.2 [4.1 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with event.

35. Secondary Outcome: Dose Expansion: Progression Free Survival (PFS) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by Blinded Independent Central Review (BICR)
Description: as for outcome 25
Time Frame: as for outcome 34
Population: FAS included all participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 19
Months | 7.2 [3.9 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with event.

36. Secondary Outcome: Dose Expansion: Overall Survival (OS): Probability of Participants Who Were Event-Free at Month 12
Description: OS was defined as the time from the first dose date to date of death due to any cause. Participant was considered as event (overall survival) free if participant was not died and was alive at Month 12. Probability of participants who were event free at Month 12 was estimated by Kaplan-Meier method and reported.
Time Frame: At Month 12
Population: as for outcome 28
Measure: Number (90% Confidence Interval); unit: Probability of event free participants
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 19
Probability of event free participants | 0.847 [0.575 to 0.951]

37. Secondary Outcome: Dose Expansion: Trough Concentrations (Ctrough) of Talazoparib
Description: Pre dose plasma drug concentration.
Time Frame: Pre dose at 0 hour on Day 1 of Cycle 2, 3, 4 and unplanned (any time during dose expansion period up to 502 days)
Population: The PK concentration analysis set included all enrolled participants who were treated and have at least 1 analyte concentration. Here "number analyzed" signifies number of participants evaluated for given time point. Data for this outcome measure was not planned to be collected and analyzed for dose escalation period, as pre-specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter
Arm/Group | Dose Expansion: Talazoparib 1.0 mg
Number analyzed (Participants) | 19
Picogram per milliliter
  Cycle 2 Day 1: number analyzed (Participants) | 12
  Cycle 2 Day 1 | 3098 (40)
  Cycle 3 Day 1: number analyzed (Participants) | 13
  Cycle 3 Day 1 | 3423 (41)
  Cycle 4 Day 1: number analyzed (Participants) | 7
  Cycle 4 Day 1 | 2910 (52)
  Unplanned: number analyzed (Participants) | 8
  Unplanned | 3670 (38)

ADVERSE EVENTS:
Time Frame: Dose escalation: maximum duration up to 286 days; Dose expansion: maximum duration up to 502 days
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety set was evaluated.
Arm/Group | Dose Escalation: Talazoparib 0.75 mg | Dose Escalation: Talazoparib 1.0 mg | Dose Expansion: Talazoparib 1.0 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 2/19
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6 | 1/19
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Talazoparib 0.75 mg (N=3) | Dose Escalation: Talazoparib 1.0 mg (N=6) | Dose Expansion: Talazoparib 1.0 mg (N=19)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Talazoparib 0.75 mg (N=3) | Dose Escalation: Talazoparib 1.0 mg (N=6) | Dose Expansion: Talazoparib 1.0 mg (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 13
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 7
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 12
Platelet count decreased (Investigations) | 0 | 2 | 6
White blood cell count decreased (Investigations) | 0 | 1 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Essential hypertension (Vascular disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 0 | 4
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail pigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 3
Malaise (General disorders) | 0 | 0 | 5
Pyrexia (General disorders) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Asthenopia (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT03343054/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03343054/SAP_001.pdf